CLINICAL TRIAL: NCT03956927
Title: Feasibility of Simulation in Therapeutic Patient Education for Adult Diabetic Patients Using the Freestyle Libre® Device
Acronym: PRE-SIMPA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: PENNECOT 2019
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Insulin-Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: Insulin-dependent diabetic patients who have participated in a full TPE program (3 sessions)
  Interventions: Other: S-TPE; Other: Questionnaires

INTERVENTIONS:
Other: S-TPE — S-TPE stimulation session with groups of 8 patients. The simulation is performed by a single patient, the others are observers in a neighbouring room where the scene is projected.
Other: Questionnaires — Pre- and post-simulation administration of self-efficacy and anxiety questionnaires (IASTA Y1 and Y2)

SUMMARY:
The benefits of Therapeutic Patient Education (TPE) have long been proven, but its implementation remains insufficient. It is only accessible to a part of the population and is too often limited to the acquisition of knowledge. TPE consists of supporting the patient in making decisions about his or her health, managing his or her life with the disease and treatment through the acquisition or maintenance of skills.

Simulation is a pedagogical method of creating fictional or reconstructed environments in order to develop skills, know-how and abilities for which direct instruction is impossible for ethical, economic or technical reasons. To date, it is recommended for the development of caregiver skills, and has been the subject of two studies among family caregivers. It seems likely that simulation will add value to the methods currently used in TPE.

To our knowledge, no studies have been conducted on simulation-based TPE (S-TPE) with patients.

A consensus conference, which is a rigorous method of comparing the opinions of experts in TPE, simulation, patient experts and caregivers, was held in order to determine the learning that could be developed through simulation and the conditions of use. However, since the patient is a specific type of learner, we hypothesize that there may be some additional conditions for the use of S-TPE. And the value of this approach remains to be demonstrated. Since the use of S-TPE has never been studied with patients, a feasibility test would make it possible to evaluate, in the context of care, the possibility of its use and its acceptance by both patients and caregivers. This is necessary before considering a multicenter trial that demonstrates an interest in developing patient skills. It was decided to carry out this study in patients with diabetes, a condition for which TPE is a precursor. Caregivers will be able to objectify the advantages and limitations of using S-TPE.

ELIGIBILITY:
Inclusion Criteria:

* Adult who has provided non-opposition to participate in the study
* Insulin-dependent diabetic patient who has participated in a complete TPE program (3 sessions) for the implementation of a FreeStyle Libre®.

Exclusion Criteria:

* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to limited judicial protection
* Pregnant, parturient or breastfeeding woman
* Adulat patients unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
level of perceived utility of the S-TPE | Through study completion, an average of 9 months
  The level of perceived utility of S-TPE for patients and caregivers through self-administered Likert scale questionnaires
Patient satisfaction: Likert scale | Through study completion, an average of 9 months
  The degree of patient satisfaction at the end of the simulation sequence by self-administered questionnaire with a Likert scale
Organizational advantages and limitations | Through study completion, an average of 9 months
  Organizational, human, material, material and temporal facilities and limitations for patients and caregivers by analyzing the verbatim of the T0 questionnaires and interviewing them at T1

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Pennecot C, Luu M, Marchand C, Gagnayre R, Dechannes N, Rudoni S, Hilaire AM, Demongeot A, Capelle D, Bardou M. First use of Simulation in Therapeutic Patient Education (S-TPE) in adults with diabetes: a pilot study. BMJ Open. 2022 Feb 28;12(2):e049454. doi: 10.1136/bmjopen-2021-049454. PMID 35228274